CLINICAL TRIAL: NCT05199116
Title: National Registry of Cardiovascular Surgery in Argentine
Acronym: ArgenCCV
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sociedad Argentina de Cardiología (Other)
Responsible Party: Sponsor
Other Study IDs: SociedadAC
Record Dates: First submitted 2020-11-06; First posted 2022-01-20 (Actual); Last update posted 2022-01-20 (Actual); Status verified 2022-01

CONDITIONS: Cardiovascular Diseases; Surgery
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The National Registry of Cardiovascular Surgery in Argentina is a registry of patients undergoing cardiovascular surgery that involves the entire country with the ultimate aim of determining the results of said surgery throughout the country.

DETAILED DESCRIPTION:
It is an observational registry with selective inclusion of patients who undergo certain cardiovascular surgeries, where the pre-surgical status will be analyzed, the determinants during surgery and the postoperative evolution of said patients will be evaluated

ELIGIBILITY:
Iinclusion Criteria:

Over 18 years

Myocardial revascularization surgery

Valvular surgeries

Ascending Aortic Surgery

Type A Aortic Dissection Surgery

Combined surgery

Exclusion Criteria:

Cardiovascular surgery for congenital pathologies

Peripheral vascular surgery

Cardiovascular surgery secondary to trauma

Thoracic and abdominal aorta pathology

Other surgeries

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients older than 18 years of age who underwent CCV according to the inclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2021-07-08 (Actual); Primary Completion 2022-08-30 (Estimated); Study Completion 2022-08-31 (Estimated)

PRIMARY OUTCOMES:
National Registry of Cardiovascular Surgery | one year
  Evaluate results of cardiovascular surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Sociedad Argentina de Cardiología, Buenos Aires, Buenos Aires F.D., Argentina

IPD SHARING:
Plan to Share IPD: Yes
the results of the registry will be analyzed by different researchers
Supporting Information: Study Protocol, SAP, ICF
Time Frame: one year

DOCUMENTS (1):
  • Study Protocol (2021-07-08): https://cdn.clinicaltrials.gov/large-docs/16/NCT05199116/Prot_000.pdf